CLINICAL TRIAL: NCT07032662
Title: A Phase 2b, Multi-center, Randomized, Double-blind, Placebo-controlled Study of IMVT-1402 Treatment in Adult Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: IMVT-1402 in Adult Participants With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMVT-1402-2401
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; IMVT-1402; Monoclonal antibody; Human immunoglobulin G1 (IgG1); CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor, care provider and outcome assessor will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMVT-1402 (Experimental)
  Interventions: Drug: IMVT-1402
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMVT-1402 — Dose 1 subcutaneous (SC) once weekly (QW) for 24 weeks (Period 1) and 52 weeks (Period 2)
  Arms: IMVT-1402
Drug: Placebo — Matching placebo SC QW for 24 weeks (Period 1)
  Arms: Placebo

SUMMARY:
This is a Phase 2b study to evaluate the efficacy and safety of IMVT-1402 in adults with CIDP.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of IMVT-1402 in adult participants with active CIDP.

ELIGIBILITY:
Inclusion Criteria:

* Have met clinical diagnostic criteria for typical CIDP or one of the following CIDP variants: multifocal CIDP or motor CIDP per the 2021 European Academy of Neurology/Peripheral Nerve Society (EAN/PNS) Guideline on Diagnosis and Treatment of CIDP.
* Have electrodiagnostic test results supporting the diagnosis of CIDP per the EAN/PNS guideline on diagnosis and treatment of CIDP.
* Are currently on, and have been receiving chronic, stable doses of systemic corticosteroids (i.e., daily or every other day oral or pulse regimen), or immunoglobulin therapy (IVIg or SCIg) ± low dose oral corticosteroids for at least 3 months for the treatment of CIDP at the time of the Screening Visit.

Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have current or prior history of IgM paraproteinemia with or without anti-myelin-associated-glycoprotein antibodies.
* Have distal, sensory, or focal CIDP, or have a diagnosis of autoimmune nodopathy per the EAN/PNS guideline on diagnosis and treatment of CIDP.
* Have polyneuropathy of causes other than CIDP including but not limited to:

  * Multifocal motor neuropathy
  * Hereditary demyelinating neuropathy
  * Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin change syndromes (i.e., POEMS)
  * Lumbosacral radiculoplexus neuropathy
  * Systemic illnesses including vitamin deficiency syndromes and paraneoplastic neuropathies
  * Drug- or toxin-induced
* Have diabetes mellitus (DM) and meets any of the following criteria:

  * Does not have both typical CIDP and strong evidence of demyelination on nerve conduction study.
  * In the opinion of the Investigator, there is evidence of poorly controlled DM preceding the diagnosis of CIDP.
  * In the opinion of the Investigator, there is evidence of poorly controlled DM at screening.
* Have a history of myelopathy or evidence of central demyelination. Additional exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants remaining Relapse-free by Week 24 | Baseline, Week 24
  Relapse is defined as a worsening (increase) of ≥ 1 point on the adjusted inflammatory neuropathy cause and treatment (aINCAT) score at any time point relative to Period 1 Baseline.

SECONDARY OUTCOMES:
Change from baseline to Week 24 in Inflammatory Rasch-Built Overall Disability Scale (I-RODS) | Baseline and Up to Week 24
Change from baseline to Week 24 in Mean Grip Strength in the dominant hand | Baseline and Up to Week 24
Change from baseline to Week 24 in Medical Research Council Sum Score (MRC-SS) | Baseline and Up to Week 24
Change from baseline to Week 24 in aINCAT score | Baseline and Up to Week 24

CONTACTS AND LOCATIONS:
Locations (134):
- United States (30):
  - Site Number - 1612, Tucson, Arizona
  - Site Number - 1618, Carlsbad, California
  - Site Number - 1619, Orange, California
  - Site Number - 1607, Rancho Mirage, California
  - Site Number -1608, San Francisco, California
  - Site Number - 1626, Parker, Colorado
  - Site Number - 1621, New Haven, Connecticut
  - Site Number - 1630, Washington D.C., District of Columbia
  - Site Number - 1601, Washington D.C., District of Columbia
  - Site Number - 1603, Maitland, Florida
  - Site Number - 1606, Miami, Florida
  - Site Number - 1617, Ormond Beach, Florida
  - Site Number - 1620, Port Charlotte, Florida
  - Site Number - 1633, Rockledge, Florida
  - Site Number - 1602, Kansas City, Kansas
  - Site Number - 1611, Nicholasville, Kentucky
  - Site Number - 1623, Boston, Massachusetts
  - Site Number - 1625, Worcester, Massachusetts
  - Site Number - 1629, Detroit, Michigan
  - Site Number - 1605, New York, New York
  - Site Number - 1627, New York, New York
  - Site Number - 1635, Chapel Hill, North Carolina
  - Site Number - 1610, Charlotte, North Carolina
  - Site Number - 1624, Canton, Ohio
  - Site Number - 1631, Yukon, Oklahoma
  - Site Number - 1614, Portland, Oregon
  - Site Number - 1616, Philadelphia, Pennsylvania
  - Site Number - 1622, Houston, Texas
  - Site Number - 1628, San Antonio, Texas
  - Site Number - 1613, Milwaukee, Wisconsin
- Argentina (4):
  - Site Number - 5002, Buenos Aires
  - Site Number - 5001, Córdoba
  - Site Number - 5003, Córdoba
  - Site Number - 5000, Rosario
- Australia (3):
  - Site Number - 5102, Brisbane
  - Site Number - 5100, Macquarie Park
  - Site Number - 5103, Parkville
- Site Number - 5200, Vienna, Austria
- Site Number - 5300, Leuven, Belgium
- Bosnia and Herzegovina (4):
  - Site Number - 5400, Banja Luka
  - Site Number - 5402, Bihać
  - Site Number - 5401, Mostar
  - Site Number - 5403, Sarajevo
- Brazil (7):
  - Site Number - 5506, Brasília
  - Site Number - 5503, Campinas
  - Site Number - 5500, Curitiba
  - Site Number - 5502, Joinville
  - Site Number - 5501, Porto Alegre
  - Site Number - 5504, Porto Alegre
  - Site Number - 5505, Vila Clementino
- Bulgaria (5):
  - Site Number - 5601, Pleven
  - Site Number - 5600, Sofia
  - Site Number - 5602, Sofia
  - Site Number - 5603, Sofia
  - Site Number - 5604, Sofia
- Site Number - 5800, Bogotá, Colombia
- Denmark (2):
  - Site Number - 3600, Copenhagen
  - Site Number - 3601, Odense
- Site Number - 7251, Tallinn, Estonia
- Site Number - 3800, Turku, Finland
- Germany (6):
  - Site Number - 6505, Berlin
  - Site Number - 6501, Bochum
  - Site Number - 6504, Essen
  - Site Number - 6500, Tübingen
  - Site Number - 6503, Ulm
  - Site Number - 6502, Würzburg
- Greece (7):
  - Site Number - 3901, Alexandroupoli
  - Site Number - 3902, Athens
  - Site Number - 3905, Chaïdári
  - Site Number - 3906, Heraklion
  - Site Number - 3903, Ioannina
  - Site Number - 3904, Larissa
  - Site Number - 3900, Pátrai
- Hungary (3):
  - Site Number - 7551, Budapest
  - Site Number - 7550, Kistarcsa
  - Site Number - 7552, Pécs
- Site Number - 4100, Waterford, Ireland
- Italy (11):
  - Site Number - 6004, Bergamo
  - Site Number - 6007, Bologna
  - Site Number - 6000, Brescia
  - Site Number - 6009, Milan
  - Site Number - 6001, Milan
  - Site Number -6005, Milan
  - Site Number - 6011, Pavia
  - Site Number - 6010, Pisa
  - Site Number - 6002, Roma
  - Site Number - 6006, Roma
  - Site Number - 6003, Siena
- Mexico (4):
  - Site Number - 2603, Colonia del Valle
  - Site Number - 2600, Culiacán
  - Site Number - 2602, Tlalpan
  - Site Number - 2601, Veracruz
- Site Number - 2200, Utrecht, Netherlands
- Site Number - 2300, Oslo, Norway
- Peru (2):
  - Site Number - 2401, Callao
  - Site Number - 2400, Lima
- Poland (9):
  - Site Number - 3007, Bydgoszcz
  - Site Number - 3008, Gdansk
  - Site Number - 3004, Katowice
  - Site Number - 3000, Krakow
  - Site Number - 3003, Krakow
  - Site Number - 3001, Lublin
  - Site Number - 3005, Lublin
  - Site Number - 3002, Poznan
  - Site Number - 3006, Warsaw
- Portugal (3):
  - Site Number -2902, Almada
  - Site Number - 2901, Matosinhos Municipality
  - Site Number - 2903, Vila Nova de Gaia
- Romania (2):
  - Site Number - 7503, Bucharest
  - Site Number - 7500, Constanța
- Serbia (4):
  - Site Number - 9000, Belgrade
  - Site Number - 9003, Belgrade
  - Site Number -9002, Kragujevac
  - Site Number - 9001, Niš
- Slovakia (3):
  - Site Number - 2800, Martin
  - Site Number - 2802, Prešov
  - Site Number - 2801, Rimavská Sobota
- Site Number - 7351, Ljubljana, Slovenia
- Spain (6):
  - Site Number - 7100, Barcelona
  - Site Number - 7101, Barcelona
  - Site Number - 7104, Bilbao
  - Site Number - 7103, Córdoba
  - Site Number - 7102, Santiago de Compostela
  - Site Number - 7105, Valencia
- Turkey (Türkiye) (6):
  - Site Number - 4250, Bakırköy
  - Site Number - 4253, Başakşehir
  - Site Number - 4255, Bursa
  - Site Number - 4251, Istanbul
  - Site Number - 4254, Izmir
  - Site Number - 4252, Samsun
- United Kingdom (4):
  - Site Number - 7001, Bristol
  - Site Number - 7002, Glasgow
  - Site Number - 7000, Salford
  - Site Number - 7003, Southampton

IPD SHARING:
Plan to Share IPD: No